CLINICAL TRIAL: NCT05916105
Title: Drug Utilization Evaluation Study of Ciprofloxacin Utilization and Adverse Events Occurrence in Community Pharmacy Setting: A Cross-Sectional Study
Brief Title: Ciprofloxacin Utilization and Adverse Events Occurrence in Community Pharmacy Setting
Status: Completed | Type: Observational
Sponsor: Damanhour University (Other)
Responsible Party: Principal Investigator, Rehab Werida, Principal Investigator, Damanhour University
Other Study IDs: Ciprofloxacin Utilization
Record Dates: First submitted 2023-06-13; First posted 2023-06-23 (Actual); Last update posted 2023-06-23 (Actual); Status verified 2023-06

CONDITIONS: Ciprofloxacin Adverse Reaction
Keywords: Ciprofloxacin; Use evaluation; Drug interaction
MeSH Terms: interventions — Ciprofloxacin

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Ciprofloxacin: 151 record of Ciprofloxacin
  Interventions: Drug: Ciprofloxacin Tablets

INTERVENTIONS:
Drug: Ciprofloxacin Tablets — Ciprofloxacin antibiotic
  Other Names: Ciprofloxacin

SUMMARY:
Background: Ciprofloxacin is a fluoroquinolone that is commonly used to treat a variety of diseases. Ciprofloxacin resistance is rising, resulting in suboptimal patient care. The goal of this study was to evaluate ciprofloxacin use in the community in terms of acceptable prescription, dose, frequency, and duration of use.

Methods: A cross-sectional research was done in Egyptian community pharmacies by community pharmacists. Patients who were administered oral ciprofloxacin during the research period were included.

DETAILED DESCRIPTION:
From September 2021 to February 2022, a cross-sectional, research was undertaken to evaluate ciprofloxacin usage. The investigation was carried out by community pharmacists in seven Egyptian community pharmacies.

Data Collection: data gathered from pharmacy patients' records on a data collection form that included the factors indicated. The General Symptoms Questionnaire, physical examination, and blood testing were used to identify adverse occurrences.

Study variables:

* age, gender, pregnancy/lactation
* Department/indication
* Dose, Frequency, Duration, Adverse events, Drug interactions.

Data was categorized and analyzed using appropriate software.

ELIGIBILITY:
Inclusion Criteria:

* All ciprofloxacin included prescription during the study period.

Exclusion Criteria:

* un included ciprofloxacin prescription.

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: A total of 151 patients' record indicated for ciprofloxacin were included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 151 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2022-03-01 (Actual)

PRIMARY OUTCOMES:
Indications | 6 months
  Appropriate Indications of ciprofloxacin (frequency )
ciprofloxacin prescription (frequency ) | 6 months
  Number of appropriate ciprofloxacin prescription
adverse events | 6 months
  adverse events occured during ciprofloxacin therapy (frequency )

CONTACTS AND LOCATIONS:
Overall Officials: Rehab H Werida, Ass. Prof., Study Director — Damanhour University
Locations (1):
- Rehab Hussein Werida, Damanhūr, Elbehairah, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Goldman MP. Ciprofloxacin drug utilization review and prospective drug use evaluation. DICP. 1990 Jan;24(1):82-6. doi: 10.1177/106002809002400115. PMID 2301191
- [Background] Davis R, Markham A, Balfour JA. Ciprofloxacin. An updated review of its pharmacology, therapeutic efficacy and tolerability. Drugs. 1996 Jun;51(6):1019-74. doi: 10.2165/00003495-199651060-00010. PMID 8736621